CLINICAL TRIAL: NCT03113981
Title: Randomized Controlled Non-inferiority Trial Assessing the Osseointegration of THA Grafted by Sodium Polystyrene Sulfonate -PolyNASS- (ACTISURF-CERAFIT® ) Versus Non-grafted THA (CERAFIT®)
Brief Title: Osseointegration of THA Grafted by PolyNASS (ACTISURF-CERAFIT® ) Versus Non-grafted THA (CERAFIT®)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Societe ACTIVBIOMAT (Industry)
Collaborators: Slb Pharma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACTISURF-OI-16; 2015-A01919-40 (Other: ID RCB - ANSM)
Record Dates: First submitted 2017-04-05; First posted 2017-04-14 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis, Hip; Coxarthrosis; Primary; Coxarthrosis; Secondary; Osteonecrosis; Aseptic, Idiopathic; Hip Arthroplasty Replacement; Hip Arthroplasty, Total; Hip Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Hip; Neoplasm Metastasis; Osteonecrosis; Infertility | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- ACTISURF-CERAFIT (Experimental): Total hip arthroplasty (CERAFIT) grafted by PolyNass
  Interventions: Device: Total Hip Arthroplasty
- CERAFIT (Active Comparator): Total hip arthroplasty (CERAFIT) with HydroxyApatite (HA) not grafted by PolyNass
  Interventions: Device: Total Hip Arthroplasty

INTERVENTIONS:
Device: Total Hip Arthroplasty — Implanting THA grafted with PolyNass or not

SUMMARY:
The infection rate after Total Hip Arthroplasty (THA) is about 1%. It is a serious condition, with high morbidity, sometimes fatal, requiring costly treatment.

The treatment is difficult because "biofilm" forms very early after the bacterial contamination of the prosthesis.

Prevent infection means reduce or prevent the formation of bacterial biofilm and controlling protein response to allow osseous-integration of the prosthesis.

A new prosthesis was developped, grafted by PolyNaSS (polysodium styrenesulfonate). This bioactive polymer allows to substantially reduce bacterial adhesion and increase biocompatibility and bio-integration in preclinical studies. This first clinical study aims to compare the osseous-integration of this prosthesis to the same prothesis with no grafting.

No previous clinical trial

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 50 and under 75 years OR aged under 50 years with joint lesions not amenable to successful conservative treatment.
* THA following a primary or secondary osteoarthritis
* THA following an aseptic osteonecrosis
* THA following a rapidly destructive osteoarthritis
* Social insurance
* Informed and signed consent

Exclusion Criteria:

* Patients younger than 50 years and with joint lesions that can be successfully treated with conservative treatment
* Inflammatory rheumatism
* Long-term corticosteroid treatment
* Tumor Pathology of the hip bone
* Study femoral stem not adapted to the patient's anatomy (verified on preoperative X-rays using Ceraver templates).
* Loss of bone of the joint that makes it impossible to properly anchor a cementless prosthesis
* Acetabular or femoral bone graft associated
* Infectious hip arthritis history
* Evolving infection of the articulation or peri-articular region involved, including severe neuroarthropathy
* Surgical history on the affected hip
* Allergy known to any component of prostheses
* Known hypersensitivity to polystyrene sulfonate resins
* Native cotyl with a diameter of less than 42mm or greater than 68mm
* Significant muscle loss, neuromuscular injury or vascular insufficiency of affected limb
* Charcot's disease
* Immunocompromised patients
* Difficulties of follow-up (departure on vacation, imminent change, geographical distance, patients not residing in metropolis, insufficient motivation) or understanding of the protocol
* Patient Refusal
* Pregnant and lactating women

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2039-12 (Estimated)

PRIMARY OUTCOMES:
Osseous-integration of the femoral stem and the acetabular component | 1 year post-surgery for both groups
  (Yes/No). THA will be judged "osseointegrated" if the acetabulum AND the femur meet the following osseous-integration criteria:
  * femur: score of Engh and Massin strictly greater than 10
  * AND acetabulum: Implant migration less than 5 mm AND no total radiolucent line and no osteocondensation at the bone-cup interface in the 3 zones of Gruen

SECONDARY OUTCOMES:
Mid-term survival rate of the hip prosthesis | 15 years post-surgery for CERAFIT group and 16 years post-surgery for ACTISURF group
  Based on the unipolar or bipolar change of the femoral head regardless of the cause, septic or mechanical.
Score ARA femur of Epinette | 1 year post-surgery for both groups
  Adaptation criteria of the bone to the cementless stem
Hip prosthesis infection rate defined according to the 2011 criteria of the Musculoskeletal Infection Society (MSIS). In case of suspicion of infection, a hip joint aspiration with synovial fluid culture will be performed. | 2 years post-surgery for both groups
  yes/no
Postel Merle d'Aubigné (PMA) score | 2 years post-surgery for both groups. 5, 10 years post-surgery for CERAFIT group. 4, 6, 8, 10, 12, 14, 16 years post-surgery for ACTISURF group.
  From 18 (perfect) to 0 (worst)
Harris Hip Score (HHS) | 2 years post-surgery for both groups. 5, 10 years post-surgery for CERAFIT group. 4, 6, 8, 10, 12, 14, 16 years post-surgery for ACTISURF group.
  10 question items and scores range from 0-100 with higher scores representing less dysfunction and better outcomes.
Forgotten Hip Score (FHS) | 2 years post-surgery for both groups. 5, 10 years post-surgery for CERAFIT group. 4, 6, 8, 10, 12, 14, 16 years post-surgery for ACTISURF group.
  12 question items and scores range from 0-100 with higher scores representing a forgotten hip (excellent)
Osseous-integration of the femoral stem and the acetabular component based on radiographies | 2 years post-surgery for both groups. 5 and 10 years post-surgery for CERAFIT group. 4, 6, 8, 10, 12, 14, 16 years post-surgery for ACTISURF group.
  Subsidence of the femoral stem, presence of periprosthetic radiolucent lines in the Gruen and Amstutz zones (femur) and in the DeLee and Charnley zones (acetabulum), Brooker score
THA survival | 6 years post-surgery for ACTISURF group. 10 years post-surgery for both groups.
  Event=THA revision (change of the stem or acetabular component) whatever the reason (infectious or mechanical failure)
Adverse and serious adverse events evaluation | For ACTISURF group: at 4, 6, 8, 10, 12, 14, 16 years post-surgery. For CERAFIT group: at 5, 10, and 15 years post-surgery.
  Occurrence of related to THA serious adverse events after 2 post-operative years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bauer, MD, PhD, Principal Investigator — Hospital Ambroise Paré Paris
Locations (7):
- France (7):
  - CHU de Bordeaux Site Pellegrin, Bordeaux
  - Hopital Ambroise Pare, Boulogne-Billancourt
  - CH Privé Brestois et Clinique Pasteur, Brest
  - CHU Cavale Blanche, Brest
  - Hôpital Lariboisière, Paris
  - CH de Cornouaille, Quimper
  - HUS, Strasbourg

IPD SHARING:
Plan to Share IPD: No